CLINICAL TRIAL: NCT04754386
Title: Caregiver-Assisted Oral Fluid-based HIV Screening in Children: Estimation of Acceptability, Feasibility and Effectiveness Linked to Index Testing Services in Zambia
Brief Title: Caregiver-Assisted Oral Fluid-based HIV Screening in Children: Zambia
Status: Completed | Type: Observational
Sponsor: Catholic Relief Services (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: CDC IRB 7272
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: HIV Testing

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Acceptability of OraQuick Advance© Rapid HIV-1/2 Antibody screening Oral fluid-based HIV test — The project offers HIV oral test kits to index parents/caregivers with children eligible for index testing services at facility settings to expand access to HIV testing and treatment services for children, and to ensure that all children who screen positive with an oral fluid-based HIV screening kit are linked to confirmatory testing, and newly diagnosed children are initiated on ART.

SUMMARY:
The purpose of this study is to evaluate the acceptability, feasibility and effectiveness of a caregiver-assisted oral fluid-based HIV test to screen children for HIV in Zambia. The results of this study are intended to support expanded access to HIV testing and treatment services for children, and to ensure that all newly diagnosed children are linked to clinical care.

DETAILED DESCRIPTION:
Rationale: Globally, there are 1.8 million children living with HIV (CLHIV); however, despite great progress over the past 15 years, only 52% are receiving antiretroviral therapy (ART), leaving approximately 864,000 children in need of treatment. According to the ZAMPHIA study, only 50.6% of HIV-positive Zambian children aged 0-14 years knew their HIV status (UNAIDS 1st 90). Pediatric case finding is the first and, critical step to close the pediatric ART gap. In Zambia, there are an estimated 25,920 CLHIV in need of HIV treatment. Reaching this population is challenging, because children are dependent on parents and caregivers to access HIV testing services. Parents and caregivers often face logistical, societal and other barriers that limit the uptake of testing services for children. In order to achieve the second and third UNAIDS 95 targets of pediatric HIV treatment coverage and viral load suppression to reach epidemic control, country programs need to utilize increasingly targeted and innovative testing modalities to optimize the identification CLHIV. Saliva-based screening tests may present a safe and reliable way to identify children living with HIV that can expand access to this essential service in resource-limited settings where most CLHIV reside.

Methods: The study will have a cross-sectional cluster sampling design, in which large facilities in two provinces will be selected using probability-proportional-to-size (PPS) sampling. Within each of 15 selected facilities, adult index parent/caregivers who are the parent/caregivers of approximately 200 children will be recruited to accept oral fluid-based HIV test kits for their children. There will be 3000 participants in the sample. Index parent/caregivers will be consented to participate in the study, given a number of OTKs corresponding to the number of children eligible for testing, followed up to confirm saliva-based test (SBT) results, participate in a testing experience survey, and return the OTK. All children screening HIV-positive will receive active linkage to confirmatory diagnostic testing, and treatment services for newly diagnosed HIV-positive children. In addition to these data, a sample (n=445) of caregivers will be asked questions regarding their experiences with administering the screening kit on their children.

ELIGIBILITY:
Inclusion Criteria for adult index parent/caregivers:

* All HIV-positive adults
* 18 years old or older with eligible children

Inclusion Criteria for Eligible children:

• All biological children (of an adult index case) 18 months - 14 years of age with an unknown HIV status

Exclusion Criteria for adult index parent/caregivers:

* Adults answering "yes" to any of the four intimate partner violence risk assessment questions
* Adults previously diagnosed as mentally disabled
* Adults currently in prison are excluded from this study.
* Adult partners of index parent/caregivers

Exclusion Criteria for Children:

* Children <18 months of age
* All biological children (of an index case) 18 months - 14 years of age with a documented HIV-negative status after cessation of breastfeeding
* All biological children (of an index case) 18 months - 14 years of age with a documented HIV-positive status
* Children still breastfeeding or with cessation of breastfeeding < 3 months
* Non-biological children of the index parent/caregiver

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At the 15 PEPFAR-supported health facilities, all eligible adult HIV-positive clients will be offered oral fluid-based HIV screening kits for their children as a part of index testing services. Study participants will be recruited during post-test counseling sessions for adults who are newly identified as HIV-positive, and/or ART clinic visits for HIV-positive adults already on treatment.
Sampling Method: Non-Probability Sample
Enrollment: 2730 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
Estimate the acceptability of implementing caregiver-assisted oral fluid-based HIV screening fluid-based HIV screening for children as a part of index testing services for index parent/caregivers. | 6 months
  * Proportion of eligible index parent/caregivers (disaggregated by sex) that accepted an oral fluid-based HIV screening kit as part of innovative index testing services for their eligible children when first offered.
  * Proportion of eligible index parent/caregivers (disaggregated by sex) that accepted an oral fluid-based HIV screening kit as part of innovative index testing services for their eligible children when they returned for a subsequent visit.
  * Proportion of eligible children (i.e. unknown HIV status) screened with an oral fluid-based HIV screening kit.
Estimate the feasibility of implementing caregiver-assisted oral fluid-based HIV screening fluid-based HIV screening for children as part of index testing services for HIV-positive adults. | 6 months
  * Proportion of index parent/caregivers who reported that the caregiver-assisted oral fluid-based HIV screening kit to screen children for HIV was easy to use.
  * Proportion of index parent/caregivers who reported needing additional assistance with administering the oral fluid-based HIV screening kit.
  * Proportion of index parent/caregivers who reported adverse events related to the use of caregiver-assisted oral fluid-based HIV screening kits to screen their children for HIV.
Estimate the effectiveness of caregiver-assisted oral fluid-based HIV screening on testing yield, return to clinic, and linkage to ART for newly identified CLHIV. | 6 months
  * Proportion of eligible children screened reactive through a caregiver-assisted oral fluid-based HIV screening kit.
  * Proportion of eligible children who screened reactive through a caregiver-assisted oral fluid-based HIV screening kit who received confirmatory testing, within 1 day, 1 week, 1 month of their reactive screen.
  * Proportion of eligible children who screened reactive through a caregiver-assisted oral fluid-based HIV screening kit who started on ART within 1 day, 1 week, 1 month of their confirmatory test.
  * Proportion of index parent/caregivers who were offered an oral fluid-based test kit to screen their eligible children for HIV used it.

SECONDARY OUTCOMES:
Estimate the cost of caregiver-assisted oral fluid-based HIV screening compared to the existing standard costs of the existing referral to testing program. | 6 months
  • Comparative costs between oral fluid-based screening and the costs of the existing referral to testing program, from the perspective of the health care provider.

CONTACTS AND LOCATIONS:
Overall Officials: Carl C Stecker, MPH, EdD, Principal Investigator — Catholic Relief Services - USCCB
Locations (15):
- Zambia (15):
  - Mutendere Clinic, Mutendere, Lusaka Province
  - Chitope Rural Health Centre, Mwavi, Lusaka Province
  - Nadezwe Rural Health Center, Chikankata, Southern Province
  - Chivuna Rural Health Centre, Livingstone, Southern Province
  - Munenga Rural Health Centre, Mazabuka, Southern Province
  - Keemba Rural Health Centre, Monze, Southern Province
  - Manungu Rural Health Centre, Monze, Southern Province
  - Chazanga Clinic, Lusaka
  - Chilanga Clinic, Lusaka
  - Chilenje Clinic, Lusaka
  - Kalingalinga Clinic, Lusaka
  - Kazimva Rural Health Clinic, Lusaka
  - Matero Clinic, Lusaka
  - Nan'gongwe Clinic, Lusaka
  - Shimabala Rural Health Centre, Lusaka

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gross J, Tumwesigye NM, Mutembo S, Moyo N, Mukose A, Chilyabanyama O, Matoba J, Parris K, Lee B, Churchill T, Williamson D, Pals S, Biribawa C, Kagaayi J, Ndubani P, Okello F, Zyambo Z, Taasi G, Magongo EN, Munthali G, Mwiya M, Nazziwa E, Awor AC, Itoh M, Boyd AM, Macleod D, Rivadeneira E, Oliver D, Ferrand RA, Stecker C; FASTER Study Team. Acceptability, feasibility, and effectiveness of caregiver-assisted HIV self-testing among children using an oral mucosal test in Uganda and Zambia: a prospective interventional study. Lancet HIV. 2025 May;12(5):e325-e337. doi: 10.1016/S2352-3018(25)00005-0. PMID 40316402